CLINICAL TRIAL: NCT01201733
Title: The Immediate Effect of Traditional Thai Massage on Brain Electrical Activity in Patients With Scapulocostal Syndrome
Brief Title: Traditional Thai Massage and Brain Electrical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Assoc Prof. Dr. Wichai Eungpinithpong, Faculty of Associated Medical Sciences, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5270900044
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2010-09

CONDITIONS: Scapulocostal Syndrome
MeSH Terms: interventions — Medicine, Thai Traditional; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Thai massage (Experimental): The participants will receive a thirty minutes session of traditional Thai massage onto the scapular region
  Interventions: Other: Traditional Thai massage
- Ultrasound therapy and hot pack (Active Comparator): The participants will receive a thirty minutes session of Ultrasound therapy and hot pack
  Interventions: Other: Ultrasound therapy and hot pack

INTERVENTIONS:
Other: Traditional Thai massage — The participants will receive a thirty minutes session of traditional Thai massage onto the scapular region
  Arms: Traditional Thai massage
Other: Ultrasound therapy and hot pack
  Arms: Ultrasound therapy and hot pack

SUMMARY:
The purpose of this study is to evaluate the immediate effect of traditional Thai massage on brain electrical activity in the patients with scapulocostal syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 50 years old
2. The participants have experienced spontaneous scapular pain (VAS ≥ 3) for longer than 12 weeks (chronic) and that at least one trigger point will be present in the scapular region (serratus posterior superior, rhomboid groups, levator scapulae and trapezius muscles). Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
3. The participants will be able to follow instructions.
4. Good communication and cooperation.

Exclusion Criteria:

1. A history of the following diseases or disorders:

   * Rotator cuff disease
   * Cervical radiculopathy
   * Degenerative shoulder joint disease
   * Shoulder stiffness
2. Contraindications of traditional Thai massage

   * Contagious skin disease
   * Injury or inflammation of muscle
   * Bone fracture and/or joint dislocation
   * Open wound
   * Uncontrolled hypertension
   * Drug and/or alcohol intoxication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG):the absolute band power in every frequency band | 1 Day
  Electroencephalography (EEG) will be assessed through the gamma,delta,theta,alpha and beta bands

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Buttagat V, Eungpinichpong W, Kaber D, Chatchawan U, Arayawichanon P. Acute effects of traditional Thai massage on electroencephalogram in patients with scapulocostal syndrome. Complement Ther Med. 2012 Aug;20(4):167-74. doi: 10.1016/j.ctim.2012.02.002. Epub 2012 Mar 2. PMID 22579427